CLINICAL TRIAL: NCT05489354
Title: Effect of a mHealth Psycho-educational Intervention (mPEI) on Self-efficacy, Coping, and Psychological Distress Among Women Receiving Chemotherapy for Breast Cancer in Nigeria: A Randomised Controlled Trial
Brief Title: mHealth Usage Among Nigeria Women Diagnosed With Breast Cancer Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Akingbade Oluwadamilare, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021.693
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Women; Psychoeducation; mHealth; Nursing; Psychological issues; Nigeria
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: The research assistants who assess outcome data, data entry and analysis will be blinded to avoid the risk of assessor bias. The assistants will not participate in any other stage of implementing the program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth psychoeducational intervention (Experimental): The intervention group will receive six weeks mHealth psychoeducational intervention (mPEI) delivered through a mobile application.
  Interventions: Other: mHealth psychoeducational intervention
- Control Group (No Intervention): No psychoeducational intervention will be given.

INTERVENTIONS:
Other: mHealth psychoeducational intervention — The mPEI program will be delivered through a mobile application (app). The app has five components which include: Breast cancer education, coping skills training, discussion forum, nurse-led consultation, and psychological support. Breast cancer education and coping skills training will be conducted by the principal investigator for 30 minutes per week for six weeks and will be delivered via text, audio and video on the mobile app. Group discussion will be moderated by the principal investigator in a text format for 30 minutes per week. Nurse-led consultation and psychological support will be provided by the oncology nurse on the research team through a 15-20-minute call in the first week, third week and fifth week.
  Arms: mHealth psychoeducational intervention

SUMMARY:
The research is studying the effect of a mHealth psychoeducational intervention on self-efficacy, coping and psychological distress of Nigerian women diagnosed with breast cancer receiving chemotherapy

The study is a two-arm assessor-blinded randomised controlled trial which will be conducted in two University Teaching Hospitals in Nigeria.

DETAILED DESCRIPTION:
Aim The study aims to develop and implement a culturally adapted mHealth psychoeducational intervention (mPEI) for Nigerian women diagnosed with breast cancer receiving chemotherapy.

Objectives

1. To evaluate the effectiveness of the programme on self-efficacy (primary outcome), coping, symptom distress, anxiety, depression, and quality of life (secondary outcomes) among women with breast cancer receiving chemotherapy
2. To explore the participants' experiences and feelings towards the intervention.

Hypothesis

It is hypothesised that participants who receive the mPEI program, when compared with the control group at baseline and immediately after the intervention, will demonstrate:

1. a significantly higher level of self-efficacy,
2. a significantly higher level of coping,
3. a significantly higher level of quality of life,
4. a significantly lower level of symptom distress,
5. a significantly lower level of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria: Include females who are:

1. newly diagnosed with breast cancer within the recent three months
2. currently receiving chemotherapy,
3. have access to a smartphone and internet,
4. are able to read and write in English,
5. are cognitively capable of completing the questionnaires,
6. consent to join the study.

Exclusion Criteria: Include females:

1. with a concurrent physical or mental illness (as these might act as a confounder)
2. cognitively impaired

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy | Pre-intervention and immediately after the six weeks intervention
  Self-efficacy for coping with cancer will be measured with the Cancer Behaviour Inventory-Brief Version (CBI-B). This is a 12-item instrument measuring confidence of individuals in performing activities that show how well they are coping with the demands of cancer and their treatment. Each item will be scored on a nine-point Likert scale with '1' meaning 'not at all confident' and '9' meaning 'totally confident'. The lowest score is 12 and the highest score is 108. Higher scores indicate greater self-efficacy in coping.

SECONDARY OUTCOMES:
Change in Coping | Pre-intervention and immediately after the six weeks intervention
  Coping will be assessed through Brief Cope Inventory. This is a 28-item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Respondents rate items on a 4-point Likert scale, ranging from 1- "I haven't been doing this at all" to 4- "I have been doing this a lot". There are 14 scales in the Brief Cope, with each measuring a specific coping strategy. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale. No items are reverse scored. High scores are indicative of psychological strength, grit, a practical approach to problem-solving and is predictive of positive outcomes.
Change in Anxiety | Pre-intervention and immediately after the six weeks intervention
  Anxiety will be assessed with the Hospital Anxiety and Depression Scale (HADS). HADS comprises anxiety and depression subscales with seven items per subscale. A total score of 0-7 is normal, 8-10 is borderline abnormal and 11-21 is abnormal.
Change in Depression | Pre-intervention and immediately after the six weeks intervention
  Depression will be assessed with the Hospital Anxiety and Depression Scale (HADS). HADS comprises anxiety and depression subscales with seven items per subscale. A total score of 0-7 is normal, 8-10 is borderline abnormal and 11-21 is abnormal.
Change in Symptom Distress | Pre-intervention and immediately after the six weeks intervention
  Symptom distress will be measured with the Monroe Dunaway (M. D.) Anderson Symptom Inventory (MDASI) which comprises 13 items to measure symptom severity and six items to measure the rate of interference of the symptoms with patient's activities of daily living. The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 NRS, with 0 being "not present" and 10 being "as bad as you can imagine." For symptom severity, there are 13 items, the highest score is 130 and the lowest is 13. Higher scores indicate higher degree of symptom severity. For symptom interference, there are six items. The highest score is 60 and the lowest score is 6. Higher scores indicate higher degree of interference of symptoms with activities of daily living.
Change in Quality of Life | Pre-intervention and immediately after the six weeks intervention
  Quality of life will be assessed using the Functional Assessment of Cancer Treatment-B (FACT-B). This instrument contains 37-items for measuring five domains of health-related quality of life in BC patients on a 5-point Likert scale. The total score for the five domains ranges from 0-148 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Ming Chow, DN, Study Chair — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (2):
- Nigeria (2):
  - Lagos State University Teaching Hospital, Lagos
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akingbade O, Hong KY, Ayo OS, Alade AS, Lawal MA, Somoye IE, Adediran V, Sado O, Chow KM. Development and feasibility of an mHealth intervention for psychoeducational support of Nigerian women diagnosed with breast cancer undergoing chemotherapy: A pilot randomized controlled trial. PLoS One. 2024 Nov 25;19(11):e0314365. doi: 10.1371/journal.pone.0314365. eCollection 2024. PMID 39585879